CLINICAL TRIAL: NCT00251433
Title: An Open-label, Multicenter, Phase I/II Dose Escalation Study of Oral GW572016 in Combination With Docetaxel (Taxotere) Plus Trastuzumab (Herceptin) in Subjects Previously Untreated for ErbB2-overexpressing Metastatic Breast Cancer
Brief Title: GW572016 With Docetaxel and Trastuzumab for the Treatment Of Untreated ErbB2 Over-Expressing Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: EGF100161 (NCT00251433) was terminated in Phase I (Phase II expansion portion of the study was never initiated) by sponsor decision.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGF100161; 2005-000846-35 (EudraCT Number); CLAP016A2101 (Other: Novartis)
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Neoplasms, Breast
Keywords: ErbB1; ErbB2; trastuzumab (Herceptin); lapatinib; Stage IV breast cancer; metastatic breast cancer; overexpression of ErbB2 receptors; docetaxel (Taxotere)
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Docetaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I (Experimental): The phase I part of the study will include cohorts of 3 patients to investigate doses of lapatinib (750mg, 1000mg, 1250mg, 1500mg) with 75mg/m2 3- weekly docetaxel plus standard weekly doses of trastuzumab with prophylactic use of growth factors in all patients. Further cohorts may be explored with prophylactic use of growth factors at the doses stipulated in the phase I dose escalation schema
  Interventions: Drug: lapatinib, docetaxel, trastuzumab

INTERVENTIONS:
Drug: lapatinib, docetaxel, trastuzumab — The phase I part of the study will include cohorts of 3 patients to investigate doses of lapatinib (750mg, 1000mg, 1250mg, 1500mg) with 75mg/m2 3- weekly docetaxel plus standard weekly doses of trastuzumab with prophylactic use of growth factors in all patients. Further cohorts may be explored with prophylactic use of growth factors at the doses stipulated in the phase I dose escalation schema
  Other Names: GW572016

SUMMARY:
This study was designed to be two-part study (Phase I/Phase II). Part I was designed to find the optimal (best) doses of GW572016, docetaxel, and trastuzumab when given together. Part II was designed to evaluate the tumor response rate (shrinkage or lack of growth) in patients receiving all three drugs compared to patients receiving only docetaxel and trastuzumab.

DETAILED DESCRIPTION:
Phase II part was cancelled before it started. Participants were only enrolled in the phase I part and NOT the phase II part.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age.

Criteria for female subjects:

* Non-child-bearing potential (i.e., women with functioning ovaries who have a current documented tubal ligation or hysterectomy, or women who are post- menopausal);
* Child-bearing potential (i.e., women with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility.) This category includes women with oligomenorrhoea (severe), women who are perimenopausal, and young women who have begun to menstruate. These subjects must have a negative serum pregnancy test at screening and agree to one of the following:
* Complete abstinence from intercourse from 2 weeks prior to administration of the first dose of study medication until 28 days after the final dose of study medication; or
* Consistent and correct use of one of the following acceptable methods of birth control:
* male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject; implants of levonorgestrel; injectable progestogen; any intrauterine device (IUD) with a documented failure rate of less than 1% per year; oral contraceptives (either combined or progestogen only); or barrier methods, including diaphragm or condom with a spermicide.
* Subjects must have an ECOG Performance Status of 0 to 1.
* Subjects must have histologically- or cytologically-confirmed invasive breast cancer with Stage IV disease.
* Subjects must have measurable lesion(s) according to RECIST criteria for phase II, however for phase I subjects evaluable disease will be allowed (including patients with bone lesion only disease).
* Prior to enrolment in the Phase I part of the study, subjects must have documentation of ErbB2 over-expression via IHC3+ or FISH+ testing. Prior to enrolment in the Phase II part of the study, subjects must have ErbB2 over-expression confirmed by a central laboratory,
* Subjects with stable CNS metastases or leptomeningeal involvement are eligible only if they are not taking oral steroids or enzyme-inducing anticonvulsants. Subjects with CNS only disease will not be allowed.
* Subjects that received prior radiotherapy must have completed radiotherapy treatment at least 4 weeks before enrolment and recovered from all treatment-related toxicities.
* Subjects must have new or archived tumour tissue available prior to study entry to evaluate levels of relevant biomarkers.
* Subjects must have a cardiac ejection fraction within the institutional range of normal as measured by Multigated Acquisition (MUGA) scan or echocardiogram (ECHO).
* Subjects must have adequate haematological, hepatic, and renal function. Haemoglobin ≥9gm/dL Absolute granulocyte count ≥1500/mm³ (1.5 x 10^9/L) Platelets ≥75,000/mm³ (75 x 10^9/L) Total bilirubin ≤1.5mg/dL Both ALT and AST ≤1.5 times the upper limit of the normal range (ULN) and alkaline phosphatase ≤2.5 times the ULN (See Taxotere Data Sheet) Serum creatinine ≤ 2.0mg/dL or calculated creatinine clearance (CrCl) ≥40mL/min according to the formula of Cockcroft and Gault
* Subjects who received a taxane as part of adjuvant or neoadjuvant therapy are eligible if they had progression of their disease more than 6 months after completion of treatment.
* Subjects who received prior ErbB inhibitors in the adjuvant setting will be allowed, but a disease-free interval of at least 6 months must be demonstrated after the end of therapy.

Exclusion Criteria:

* Subject has peripheral neuropathy of grade 2 or higher;
* Subject has had prior systemic therapy (except one line of hormonal therapy) for metastatic disease. Also, any subjects with prior chemotherapy in the adjuvant or neoadjuvant setting with anthracycline or anthracenedione-containing regimens with cumulative doses of ≥360mg/m² of doxorubicin, ≥720mg/m² of epirubicin, or ≥72mg/m² of mitoxantrone;
* Subjects with prior systemic investigational drugs within the past 30 days or topical investigational drugs within the past 7 days;
* Subjects with uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure;
* Subjects with a known immediate or delayed hypersensitivity or untoward reaction to docetaxel, trastuzumab, or other related compounds, or to drugs chemically related to lapatinib. These include other aminoquinazolines, such as gefitinib (Iressa), erlotinib (Tarceva), or other chemically-related compounds.
* Subjects taking any prohibited medications
* Subject neither affiliated with, nor beneficiary of a social security category (For France only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-09-26 (Actual); Primary Completion 2010-06-10 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Phase I: Optimal doses and toleration of the three drugs administered together. | 3 weeks
Phase II: The primary efficacy endpoint is objective tumour response rate as measured by radiological imaging, photography, and/or physical examination performed every other cycle and recorded according to RECIST criteria. | 3 weeks

SECONDARY OUTCOMES:
Phase I and II Tumor response rate; Time to tumor response; Length of response; Time to progression of cancer; Overall survival. | 6 weeks
PK endpoints: Cmin and Cmax; Concentrations of alpha-1 acid glycoprotein and albumin. | 6 weeks
Safety and tolerability endpoints will consist of evaluation of AEs and changes from baseline in laboratory values. | 6 weeks
Relevant biomarkers, including ErbB1, ErbB2, ErbB3, ErbB4, AKT, and potentially other biomarkers downstream from the ErbB1 and ErbB2 receptors, will be determined from tumour tissue. | 6 weeks
Serum concentrations of ErbB1 and ErbB2 ECD will be correlated to tumour response. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Nashville, Tennessee, United States
- Novartis Investigative Site, Paris, France
- Novartis Investigative Site, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Crown J, Kennedy MJ, Tresca P, Marty M, Espie M, Burris HA, DeSilvio M, Lau MR, Kothari D, Koch KM, Dieras V. Optimally tolerated dose of lapatinib in combination with docetaxel plus trastuzumab in first-line treatment of HER2-positive metastatic breast cancer. Ann Oncol. 2013 Aug;24(8):2005-11. doi: 10.1093/annonc/mdt222. PMID 23878115
- See also: Related Info — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18028